CLINICAL TRIAL: NCT06048666
Title: Effect of Intra-ovarian Injection of Autologous Platelet Rich Plasma on Ovarian Reserve Parameters and Intra Cytoplasmic Sperm Injection Outcomes in Patients With Diminished Ovarian Reserve
Brief Title: Platelet Rich Plasma on Ovarian Reserve Parameters and Intra Cytoplasmic Sperm Injection Outcomes in Patients With Diminished Ovarian Reserve
Status: Unknown | Phase: Phase 3 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Beni-Suef University (Other)
Responsible Party: Principal Investigator, Sara Abdallah Mohamed Salem, principle investigator/Lecturer of Gynecology and obstetrics Faculty of medicine Beni-Suef University, Beni-Suef University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: PRP in poor ovarian reserve
Record Dates: First submitted 2023-09-16; First posted 2023-09-21 (Actual); Last update posted 2023-09-21 (Actual); Status verified 2023-09

CONDITIONS: IVF
Keywords: platelet rich plasma , poor ovarian reserve

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intra ovarian by platelet rich plasma (Experimental): intra-ovarian injection of autologous platelet rich plasma 3 months after the PRP injection,they will undergo assisted reproductive therapy with antagonist protocol followed by a dose of 450 units of FSH (Gonal F)
  Interventions: Biological: Intra ovarian by platelet rich plasma
- control (No Intervention): they will undergo ICSI trial with antagonist protocol followed by a dose of 450 units of FSH (Gonal F)

INTERVENTIONS:
Biological: Intra ovarian by platelet rich plasma — On the day of PRP infusion (within 10 days after completion of menstrual bleeding) we will take 20 cc of venous blood from each participant of group A to prepare PRP. The blood will be transferred to a tube containing sodium citrate and centrifuged at 800 RPM for 15 min and 2000 RPM for 5 min in two stages, respectively. Then, by discarding part of the plasma, PRP will be prepared with a final concentration of one million platelets per microliter. The PRP will be injected into the ovary under spinal anesthesia and a transvaginal ultrasound guide.
  Arms: Intra ovarian by platelet rich plasma

SUMMARY:
The aim of this study is to evaluate the efficacy of intra ovarian injection of autologous platelet rich plasma on ovarian reserve parameters and ICSI outcomes in poor ovarian reserve.

DETAILED DESCRIPTION:
fifty_six infertile women suffering from poor ovarian reserve &following up at IVF Unit of Beni_suef University hospital. , and they fulfilled inclusion and exclusion criteria. they will be classlfied into two groups: Group A (study group) (involve 28 patient ):will be injected intra ovarian by platelet rich plasma Group B (control group) (involve 28 patient): will not be injected intra ovarian by platelet rich Plasma

The researcher will introduce himself to all participants included in this study and requested that they participate after explaining the purpose of the study. All participants will be given detailed information about the study's goal and predicted advantages. All participants will give their informed verbal agreement, and the data will be kept confidential. All patients will be subjected to:

Complete history was taken with special emphasis on:

Personal ,past,family&surgical history. Menstrual historyObstetric history

Clinical examination:

Physical examination included General examination: Weight, Height, BMI, Abdominal examination , Local (Pelvic) examination

Ultrasound examination:

The women will be in lithotomy position with an empty bladder. On day 2 of the menstrual cycle or withdrawal bleed, a sterile vaginal speculum has been introduced, and a TV ultrasonography probe (7.0-MH endo-vaginal probe) has been placed in the vagina roughly 1 cm away from the cervix to evaluate the volume of the ovary and antral follicle counts (AFC).

Investigations:

General (CBC, urinalysis, Random blood sugar) when needed. Specific: Hormonal profile in all patients of the study, the following were obtained prior to the procedure: Anti-Mullerian hormone (AMH). FSH, Estradiol.

* PRP preparation and time of injection On the day of PRP infusion (within 10 days after completion of menstrual bleeding) we will take 20 cc of venous blood from each participant of group A to prepare PRP. The blood will be transferred to a tube containing sodium citrate and centrifuged at 800 RPM for 15 min and 2000 RPM for 5 min in two stages, respectively. Then, by discarding part of the plasma, PRP will be prepared with a final concentration of one million platelets per microliter. The PRP will be injected into the ovary under spinal anesthesia and a transvaginal ultrasound guide.
* Patien assessment and Follow up. patients injected with PRP will be managed expectantly for 6 weeks to allow spontaneous pregnancy, at the beginning of second menstrual cycle AMH, FSH, AFC will be reassessed.
* 3months after the PRP injection, all women considered poor responders (2groups)will undergo assisted reproductive therapy with antagonist protocol followed by a dose of 450 units of FSH (Gonal F, CinnaGen, Iran). Six days after gonadotropin therapy, vaginal ultrasound will be performed to measure follicle diameter. Once the follicular size is 12 mm, the GnRH antagonist (Cetrorelix, Merck-Serono, Germany) will begin, and gonadotropin continued. When at least two dominant follicles reach the diameter of 18 mm on ultrasound, ovulation will be stimulated using 10,000 units of HCG, and oocyte retrieval will be performed under general anesthesia 34 to 36 h after the HCG injection and the two groups will be compared in terms of the outcomes such as duration of stimulation dosage of gonadotrophine serum of estradiol level on the triggering day ,number and quality of oocytes and embryons and clinical pregnancy

ELIGIBILITY:
Inclusion Criteria:

* Women under the age of 40.
* have been infertile for more than a year
* have had at least one previous unsuccessful (or cancelled) IVF cycle.
* having one of the criteria of poor ovarian response including anti mullerian hormone (AMH) level <1.1 ng /ml ,the antral follicle count of two ovaries in vaginal ultrasound <7 .

Exclusion Criteria:

* pregnancy(ruled out and documented before PRP injection) . Hydrosalpinex,uterine malformations and abnormal uterine cavity.
* Partner with severe male factor
* Ongoing malignancy.
* Chronic pelvic pain
* A history of major lower abdomen surgeries that resulted in pelvic adhesions.

Ages: 20 Years to 45 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 56 (Estimated)
Dates: Start 2023-10-30 (Estimated); Primary Completion 2024-03-30 (Estimated); Study Completion 2024-09-30 (Estimated)

PRIMARY OUTCOMES:
number of retrieved oocytes | 1 month of induction for ICSI trial
  number of oocytes obtained in ovum pick up

CONTACTS AND LOCATIONS:
Locations (1):
- Beni-suef university Hospital, Banī Suwayf, Beni Suweif Governorate, Egypt

IPD SHARING:
Plan to Share IPD: Undecided